CLINICAL TRIAL: NCT07405502
Title: The Effect of Transcutaneous Electrical Nerve Stimulation on Pain, Nausea, Vomiting, and Quality of Recovery in Patients After Retrograde Intrarenal Surgery: A Randomized Controlled Trial
Brief Title: The Effect of Transcutaneous Electrical Nerve Stimulation in Patients After Retrograde Intrarenal Surgery
Acronym: RIRS TENS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Collaborators: The Scientific Research Project Fund of Yozgat Bozok University (Unknown)
Responsible Party: Principal Investigator, Ozlem Sahin Akboga, Asist. Prof., Bozok University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Yozgat Bozok Univercity; SRPC (Other: Yozgat Bozok University Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2026-01-21; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Urinary Calculus
Keywords: Transcutaneous Electrical Nerve Stimulation; Retrograde Intrarenal Surgery; Quality of Recovery
MeSH Terms: conditions — Urinary Calculi | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: This study employs a prospective, randomized, controlled, two-arm intervention model. Eligible participants will be randomly assigned to either the TENS intervention group or the control group using a simple randomization method. The intervention group will receive standardized TENS applications during the first 24 hours postoperatively in addition to routine postoperative care, while the control group will receive routine care only. Outcome measures, including pain intensity, frequency of nausea and vomiting, and quality of recovery, will be assessed at predefined time points using validated measurement scales by blinded assessors to minimize bias. Data will be analyzed comparatively between groups to determine the effectiveness of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS group (Experimental): Intervention Arm (TENS Group): Participants in this arm will receive Transcutaneous Electrical Nerve Stimulation (TENS) in addition to standard postoperative care following Retrograde Intrarenal Surgery (RIRS). TENS will be applied using surface electrodes placed on the appropriate dermatomal areas related to the surgical site. The stimulation parameters (frequency, intensity, and duration) will be standardized for all participants and administered within the first 24 hours postoperatively. The intervention aims to reduce postoperative pain, as well as the frequency of nausea and vomiting, and to improve overall quality of recovery.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation
- Control Arm (No Intervention): Control Arm (Standard Care Group): Participants in this arm will receive standard postoperative care only, without any TENS application. Standard care will include routine monitoring, prescribed analgesic and antiemetic medications as needed, mobilization, and nursing care according to institutional protocols. Outcomes related to pain, nausea, vomiting, and quality of recovery will be assessed at the same time points as in the intervention arm to allow for valid comparison between groups.

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation — This intervention is distinguished by the early, standardized, and nonpharmacological application of Transcutaneous Electrical Nerve Stimulation (TENS) within the first 24 hours following Retrograde Intrarenal Surgery (RIRS). Unlike conventional postoperative management that primarily relies on pharmacological analgesics and antiemetics, this approach emphasizes a nurse-administered, bedside, and patient-centered neuromodulation technique that is integrated into routine care without adding invasive procedures. The use of uniform stimulation parameters, predefined electrode placement protocols, and blinded outcome assessment ensures consistency and methodological rigor, allowing the specific effects of TENS on postoperative pain, nausea, vomiting, and quality of recovery to be isolated and compared reliably against standard care.
  Arms: TENS group

SUMMARY:
This study is designed to evaluate the effects of Transcutaneous Electrical Nerve Stimulation (TENS) on pain, nausea, vomiting, and quality of recovery in patients undergoing Retrograde Intrarenal Surgery (RIRS). This prospective, randomized controlled trial, designed as a two-group study, will be conducted at the Department of Urology, Yozgat Bozok University Health Practice and Research Center between September 2025 and September 2026. A total of 72 patients who underwent RIRC and met the inclusion criteria will be included in the study. Participants will be randomly divided into two groups: an intervention group receiving TENS (n=36) and a control group without TENS (n=36). Pain levels, frequency of nausea and vomiting, and quality of recovery in both groups will be compared within the first 24 hours postoperatively. This study is expected to provide evidence-based data on the effectiveness of TENS, a non-pharmacological method, in symptom management after RIRS.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have undergone RIRS will be included in our study. Eligibility criteria include being between 18 and 70 years of age,
* Participants having an American Society of Anesthesiologists (ASA) physical status classification of I or II,
* Participants must have sufficient cognitive function and language skills to proceed with the study.

Exclusion Criteria:

* Exclusion criteria include the presence of a painful condition (e.g., inflammatory rheumatic disease, lumbar muscle degeneration, lumbar disc protrusion with back pain, acute or chronic nephritis, and pyelonephritis),
* Major organ system disease,
* Participants with pacemakers,
* Participants using analgesic medications or those with a history of significant drug abuse,
* Those with uncontrolled hypertension, diabetes or malignancies, a history of epilepsy, pregnancy, and breastfeeding,
* Participants in other clinical trials will also be excluded (Mora et al., 2007; Tu et al., 2019).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure (postoperative pain intensity) | 0-24 hours postoperatively
  The primary outcome of this study is the intensity of postoperative pain within the first 24 hours following retrograde intrarenal surgery (RIRS). Pain level will be assessed using the validated and reliable Numerical Rating Scale (NRS).
  Scale Description:
  Scale name: Numerical Rating Scale (NRS) Minimum value: 0 (no pain) Maximum value: 10 (unbearable pain) Higher score: Indicates a worse clinical outcome Unit of Measure: Scale total score

SECONDARY OUTCOMES:
Postoperative Nausea and Vomiting (PONV) Intensity Scale | 0-24 hours postoperatively
  The frequency and severity of nausea and vomiting occurring within the first 24 hours after surgery will be assessed and recorded using the Postoperative Nausea and Vomiting (PONV) Intensity Scale.
  Scale Description:
  Scale name: Postoperative Nausea and Vomiting (PONV) Intensity Scale Minimum value: 0 (no nausea/vomiting) Maximum value: 4 (severe and persistent nausea/vomiting) Higher score: Indicates a worse clinical outcome Unit of Measure: Scale total score
Quality of recovery | 24 hours postoperatively
  The quality of postoperative recovery will be assessed using the Quality of Recovery-15 Questionnaire (QoR-15), which has proven validity and reliability.
  Scale Description:
  Scale name: Quality of Recovery-15 (QoR-15) Minimum value: 0 Maximum value: 150 Higher score: Indicates better recovery quality Unit of Measure: Scale total score

OTHER OUTCOMES:
Analgesic and antiemetic consumption | Post-surgery 0-24 hours
  Total doses of analgesic and antiemetic drugs administered within the first 24 hours post-surgery (in units/day) will be calculated from patient records. The average numbers obtained for both groups will be compared.
  Unit of Measure: Pharmacological consumption amount/number (units/day)
Antiemetic Consumption | 0-24 hours postoperatively
  Description: Total antiemetic drug consumption within the first 24 hours after surgery will be extracted from medical records.
  Unit of Measure: Total dose (units/day)
Time to First Mobilization | Within 24 hours postoperatively
  Description: Time from completion of surgery to first ambulation will be recorded under standardized clinical conditions.
  Unit of Measure: Minutes
Patient Satisfaction with Postoperative Care | 24 hours postoperatively
  Description: Patient satisfaction with postoperative care will be assessed using a 0-10 Numerical Rating Scale (NRS), where higher scores indicate greater satisfaction.
  Unit of Measure: Scale total score (0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Yozgat Bozok Univercity, Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) generated in this study-including demographic characteristics, baseline clinical variables, intervention allocation, outcome measures (pain scores, nausea and vomiting frequency, quality of recovery scores), and related metadata-will be made available upon reasonable request. Data will be shared with academic institutions, regulatory bodies, or scientific journals for purposes of verification, secondary analysis, or publication requirements, subject to approval by the study's ethics committee and the execution of a data use agreement to ensure confidentiality, ethical use, and compliance with applicable data protection regulations.
Supporting Information: SAP
Time Frame: January 2026-December 2027
Access Criteria: De-identified individual participant data (IPD) generated in this study-including demographic characteristics, baseline clinical variables, intervention allocation, outcome measures (pain scores, nausea and vomiting frequency, quality of recovery scores), and related metadata-will be made available upon reasonable request. Data will be shared with academic institutions, regulatory bodies, or scientific journals for purposes of verification, secondary analysis, or publication requirements, subject to approval by the study's ethics committee and the execution of a data use agreement to ensure confidentiality, ethical use, and compliance with applicable data protection regulations.

REFERENCES:
- [Background] Kim, H. Y., Park, J. H., & Yoon, H. J. (2020). The effects of transcutaneous electrical nerve stimulation on postoperative pain and recovery in patients undergoing urological surgery: A randomized controlled trial. Journal of Urology and Renal Diseases, 5(2), 1035-1041. https://doi.org/10.23880/oajurd-16000201